CLINICAL TRIAL: NCT02915393
Title: System Biology Research of Spleen Qi Deficiency Associated "Qi Deficiency Constitution-Disease"
Brief Title: System Biology of Spleen Deficiency Syndrome
Acronym: SBSDS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Anlong Xu, President, Beijing University of Chinese Medicine
Other Study IDs: 81430099
Record Dates: First submitted 2016-09-17; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Gastritis, Atrophic; Gastric Cancer
Keywords: Chronic Gastritis; Qi Deficiency Constitution; Next Generation Sequencing; Proteomics; Metabonomics
MeSH Terms: conditions — Gastritis, Atrophic; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — frozen tissue, whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (9):
- Healthy Volunteers (BC): Healthy Volunteers with Balanced Constitution(n=10).
- Healthy Volunteers(QC): Healthy Volunteers with Qi Deficiency Constitution(n=10).
- Healthy Volunteers(DC): Healthy Volunteers with Damp-heat Constitution(n=10).
- Superficial Gastritis(SDS): Superficial Gastritis with Spleen-qi Deficiency Syndrome(n=10).
- Superficial Gastritis(DS): Superficial Gastritis with Damp-heat Syndrome(n=10).
- Atrophic Gastritis(SDS): Atrophic Gastritis with Spleen-qi Deficiency Syndrome(n=10).
- Atrophic Gastritis(DS): Atrophic Gastritis with Damp-heat Syndrome(n=10).
- Gastric Cancer(SDS): Gastric Cancer with Spleen-qi Deficiency Syndrome(n=10).
- Gastric Cancer(DS): Gastric Cancer with Damp-heat Syndrome(n=10).

SUMMARY:
Spleen Deficiency Syndrome(SDS)is a widely researched issue, but due to the limitations of the research methods, the scientific mechanism of SDS is biased and not comprehensive. SDS would be researched in this project deeply and systematically with modern life-scientific methods. Based on the previous work, the participants, with SDS, suffering from Qi deficiency syndrome--chronic superficial gastritis--chronic atrophic gastritis--gastric cancer would be included, and the corresponding research would be conducted at the molecular-cell-gastric tissue level, and at the same time, systematical biological database of SDS would be built by systematical biological methods, such as pioneered SPARS sequencing technology created in our research group, proteomics and metabonomics. Under the above work, the investigators would conduct data mining and molecular network analysis, and then verify the key functions. By analyzing the systematical biological features of syndrome and its relationships with constitution and disease, this study would provide a new basis for objective reality of syndrome, and also offer a crucial premise of revealing biological basis for syndrome correctly, which is of important theoretical and practical significance.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years.
* No apparent abnormality in the routine blood test, urinalysis, routine stool & fecal occult blood test, biochemical test, chest radiograph and electrocardiogram(ECG).
* The endoscopic diagnoses of chronic superficial gastritis, chronic atrophic gastritis and gastric cancer conform to the corresponding pathological diagnoses
* TCM diagnoses of Spleen-qi Deficiency Syndrome or Spleen Damp-heat Syndrome.
* Voluntary participation.
* Having given written informed consent.

Exclusion Criteria:

* Gastropathy with special causes, such as acute gastritis, gastrinoma, chronic gastritis resulting from special causes (like granulomatous gastritis, lymphocytic gastritis, eosinophilic gastritis, gastritis after gastric operation) peptic ulcer, other malignant tumors of stomach (like gastric lymphoma, gastri stromal tumor, carcinoid tumor, malignant hemangioma, squamous-cell carcinoma, primary gastric choriocarcinoma and metastatic gastric tumor), benign gastritic tumors that originate from epithelium or submucosa (epithelial tumors like adenomatous polyps and hyperplastic polyps, stromal tumors like benign stromal tumor, neuronal tumor and pseudolymphoma).
* Combined with other digestive diseases (like gastroesophageal reflux, esophageal varices, acute and chronic hepatitis and cirrhosis arising from various causes, acute/chronic pancreatitis and acute/chronic cholecystitis).
* Combined with other severe systemic diseases such as respiratory failure, severe cardiovascular and cerebrovascular, immune system, urinary and mental disorders diseases.
* Pregnancy, or planning pregnancy during the trial or within three month period thereafter.
* Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 90 cases will be gathered between August, 2016 and September, 2017. All the cases include: ①10 healthy volunteers in Beijing with balanced constitution, 10 with Qi Deficient Constitution (Spleen-qi Deficiency Syndrome) and 10 with Damp-heat Constitution. ②Patients in Dongfang Hospital diagnosed as chronic superficial gastritis,chronic atrophic gastritis or gastric cancer, 20 for each disease and half of each with Spleen-qi Deficiency Syndrome, half with Spleen Damp-heat Syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Examination of the stomach with an endoscope. | at the beginning of the enrollment
  Endoscopic diagnosis standard of chronic gastritis according to Chinese Society of Digestive Endoscopy.
Pathological biopsy of gastric mucosa. | at the beginning of the enrollment
  Pathological diagnosis standard of chronic gastritis according to Chinese Society of Gastroenterology.Pathological diagnosis standard of gastric cancer according to Ministry of Health P.R.China
Detection of helicobacter pylori by Urea Breath Test(UBT) | at the beginning of the enrollment

SECONDARY OUTCOMES:
Analysis of gastric mucosa/venous blood/urine by system biology techniques | Three measurements within 1 year
Constitutional classification of TCM assessed by the Traditional Chinese Medicine Physical Constitution Scale | at the beginning of the enrollment
TCM syndrome type diagnosed by two professional TCM doctors | at the beginning of the enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Anlong Xu, Principal Investigator — Beijing University of Chinese Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] You L, Zhang S, Li T, Sang X, Li K, Wang W, Gao X, Wu J, Huang G, Wang T, Xu A. Integrated analyses of miRNA and mRNA profiles in leukocytes and serums in traditional Chinese medicine (TCM)-defined Pi-qi-deficiency syndrome and Pi-wei damp-heat syndrome resulting from chronic atrophic gastritis. Chin Med. 2021 Jan 6;16(1):4. doi: 10.1186/s13020-020-00416-9. PMID 33407671